CLINICAL TRIAL: NCT03822793
Title: Dose Study of Tranexamic Acid in Total Hip Replacement to Reduce Post-operative Hemoglobin Loss: A Phase 2 Randomized Double-blind Monocentric Study
Brief Title: A Dose-response Study of Tranexamic Acid in Total Hip Arthroplasty
Acronym: PRADO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18CH052; 2018-004552-37 (EudraCT Number); 2022-502532-38-01 (Other: CTIS)
Record Dates: First submitted 2018-12-31; First posted 2019-01-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Arthropathy of Hip
Keywords: tranexamic acid (TXA); arthroplasty; hip; Exacyl
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomized double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Patient will be included in this group by randomization and they will receive an intravenous perfusion of NaCl (sodium chloride 9%; placebo) intravenous over 9 minutes, starting at the time of surgical incision.
  Interventions: Drug: Placebo
- Group 1: perfusion of 300 mg Exacyl (Experimental): Patient will be included in the group 2 by randomization and they will receive an intravenous perfusion of 300 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Interventions: Drug: Group 1: perfusion of 300 mg Exacyl
- Group 2: perfusion of 500 mg Exacyl (Experimental): Patient will be included in the group 2 by randomization and they will receive an intravenous perfusion of 500 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision..
  Interventions: Drug: Group 2: perfusion of 500 mg Exacyl
- Group 3: perfusion of 1000 mg Exacyl (Experimental): Patient will be included in the group 3 by randomization and they will receive an intravenous perfusion of 1000 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Interventions: Drug: Group 3: perfusion of 1000 mg Exacyl
- Group 4: perfusion of 3000 mg Exacyl (Experimental): Patient will be included in the group 4 by randomization and they will receive an intravenous perfusion of 3000 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Interventions: Drug: Group 4: perfusion of 3000 mg Exacyl

INTERVENTIONS:
Drug: Placebo — Patient will receive an intravenous perfusion of NaCl (sodium chloride 9%; placebo) intravenous over 9 minutes, starting at the time of surgical incision.
  Arms: Placebo
Drug: Group 1: perfusion of 300 mg Exacyl — Patient will receive an intravenous perfusion of 300 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Arms: Group 1: perfusion of 300 mg Exacyl
Drug: Group 2: perfusion of 500 mg Exacyl — Patient will receive an intravenous perfusion of 500 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Arms: Group 2: perfusion of 500 mg Exacyl
Drug: Group 3: perfusion of 1000 mg Exacyl — Patient will receive an intravenous perfusion of 1000 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Arms: Group 3: perfusion of 1000 mg Exacyl
Drug: Group 4: perfusion of 3000 mg Exacyl — Patient will receive an intravenous perfusion of 3000 mg Exacyl (tranexamic acid) intravenous (IV) over 9 minutes, starting at the time of surgical incision.
  Arms: Group 4: perfusion of 3000 mg Exacyl

SUMMARY:
A single preoperative dose of tranexamic acid (TXA) reduces blood loss and red blood cell transfusion in primary hip arthroplasty. Numerous regimens have been tested, ranging from 10mg/kg up to 3g. However the optimal dose to administer is unknown.

DETAILED DESCRIPTION:
This dose-response study is a randomized double blind study with five groups of 30 patients each. Patients will be randomized to placebo, tranexamic acid (TXA) 300 mg, tranexamic acid (TXA) 500 mg, tranexamic acid (TXA) 1000 mg or tranexamic acid (TXA) 3000 mg. In addition a pharmacokinetic/pharmacodynamic study will be performed to identify the contribution of tranexamic acid (TXA) plasma concentration as a predictor of intra and postoperative D-Dimer values.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring primary hip arthroplasty (less than 3 months)
* Informed Consent from the patient or their legally authorized representative
* Affiliation to French Social Security Healthcare system

Exclusion Criteria:

* Hip fracture of less than 3 months
* Bilateral hip arthroplasty or anterior approach to hip arthroplasty
* Haemorrhagic surgery in the previous 2 weeks
* Contraindication to tranexamic acid
* Contraindication to apixaban
* Chronic use of anticoagulant
* Pregnancy
* Previous participation to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
haemoglobin decrease in the perioperative period | Day 1 to Day 4
  Percentage of haemoglobin change in the perioperative period. It requires the sampling of haemoglobin just before surgery (Day 1) and on the fourth postoperative day

SECONDARY OUTCOMES:
Tranexamic acid pharmacokinetics | Day 1
  For tranexamic acid pharmacokinetics, the outcome measure is the sampling of tranexamic blood concentration.
D-Dimer kinetics | Day 1
  For tranexamic acid pharmacodynamics, the outcome is the sampling of D-Dimer levels.
allogenic red blood cell transfusion | Day 1 to day 8
  For allogenic red blood cell transfusion, the outcome measure will be the percentage of patients that will receive the transfusion of at least one allogenic red blood cell unit in the perioperative period.
severe anaemia | Day 1 to day 8
  For severe anaemia (defined as a level of haemoglobin <10 gram by deciliter), the outcome measure will be the percentage of patients that will have at least one value of haemoglobin <10 gram by deciliter in the perioperative period.
incidence of symptomatic thrombotic events and death | Day 1 to day 8
  For the incidence of symptomatic thrombotic events and death, the outcome measure is a combined criteria of venous events (deep venous thrombosis or pulmonary embolism), arterial events (acute coronary syndrome, stroke or peripheral arterial thrombosis) and death.
occurrence of a seizure | Day 8
  The endpoint is a combined criteria endpoint involving either the clinical observation of a generalized tonic-clonic seizure or a partial seizure or an epilepsy confirmed by an electroencephalogram interpreted by a neurologist blinded to the patient's inclusion group.
number of adverse events | Day: 45
  collection in medical records the adverse events at 45 days after surgery :
  * venous thrombo-embolism / arterial
  * hematoma leading to modification of rehabilitation or requiring revision surgery
  * infections of superficial or deep surgical site

CONTACTS AND LOCATIONS:
Overall Officials: Julien LANOISELEE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zufferey PJ, Barrat E, Deygas B, Lanoiselee J, Ollier E. Dose-effect relationship of intravenous tranexamic acid on perioperative haemoglobin drop in total hip arthroplasty (PRADO study): study protocol for a randomised, double-blind, placebo-controlled, dose-response study. BMJ Open. 2025 Dec 3;15(12):e100265. doi: 10.1136/bmjopen-2025-100265. PMID 41338640